CLINICAL TRIAL: NCT05820867
Title: Prospective Comparison of Single vs. Staged Extractions: OHRQoL Outcomes for Wisdom Teeth Removal
Brief Title: Comparing OHRQoL: One or Two Sessions for Wisdom Teeth Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUDHF_FB_005
Record Dates: First submitted 2023-03-25; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Impacted Third Molar Tooth; Impacted Tooth
Keywords: Quality of Life; Oral health; Prospective Studies; Molar, Third; Tooth Extraction; Patient Preference
MeSH Terms: conditions — Tooth, Impacted; Patient Preference

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-session arm (Active Comparator)
  Interventions: Procedure: Single-Session Bilateral Mandibular Third Molar Extraction
- Two-session arm (Active Comparator)
  Interventions: Procedure: Two-Session Bilateral Mandibular Third Molar Extraction

INTERVENTIONS:
Procedure: Single-Session Bilateral Mandibular Third Molar Extraction — Participants in this group chose to have both of their lower mandibular third molars extracted during a single appointment. This group will be used to compare the impact of single-session extraction on patients' oral health-related quality of life, postoperative pain, and maximum interincisal opening.
  Arms: Single-session arm
Procedure: Two-Session Bilateral Mandibular Third Molar Extraction — Participants in this group chose to have their lower mandibular third molars extracted during two separate appointments. This group will be used to compare the impact of two-session extraction on patients' oral health-related quality of life, postoperative pain, and maximum interincisal opening.
  Arms: Two-session arm

SUMMARY:
This single-center prospective cohort study includes patients aged 18-30 years aimed to compare the effects of bilateral extraction of wisdom teeth at a single appointment (Group A) versus two separate appointments (Group B) on patients' oral health-related quality of life (OHRQoL). The primary outcome is Oral Health Impact Profile 14 score, while secondary outcomes included postoperative pain and maximum interincisal opening.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the Oral and Maxillofacial Surgery Department for bilateral extraction of impacted mandibular third molars.
* Asymptomatic, impacted mandibular third molars.
* Impaction classified as Class I, Position A according to the Pell and Gregory classification.
* Patients with an ASA (American Society of Anesthesiologists) Physical Status Classification of ASA 1.

Exclusion Criteria:

* Local pathology associated with third molars (e.g., cysts or tumors).
* Diagnosis of acute pericoronitis.
* Usage of anti-inflammatory drugs or antibiotics within the last week.
* Operations requiring osteotomy.
* Patients with psychiatric disorders or taking drugs that may impair their mental health.
* Patients unwilling to undergo data collection procedures.
* Pregnant or lactating women.
* Heavy smokers.
* Operations lasting longer than 45 minutes for one side (from the time the first incision is made to the last suture placed).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline oral health-related quality of life at 14 days | Baseline, postoperative day 2, day 3, day 7, day 9, and day 14
  The Oral Health Impact Profile-14 (OHIP-14) questionnaire is used to evaluate the participants' oral health-related quality of life. The OHIP-14 is a validated instrument that assesses the perceived impact of oral conditions on an individual's well-being across 14 items, each scored on a 5-point Likert scale. Lower scores indicate better OHRQoL.

SECONDARY OUTCOMES:
Change from baseline postoperative pain at 14 days | Postoperative 6th hour, 12th hour, day 2, day 3, day 7, day 9, and day 14
  The Visual Analog Scale (VAS) is used to assess the intensity of postoperative pain experienced by participants. The VAS is a validated tool consisting of a horizontal or vertical line, usually 100 mm in length, with anchor points of "no pain" at one end and "worst imaginable pain" at the other. Participants are asked to mark the point on the line that corresponds to their pain level. Higher scores indicate greater pain intensity.
Change in maximum interincisal opening | Baseline and postoperative day 7
  Maximum interincisal opening (MIO) is being measured to evaluate trismus, or restricted mouth opening, following the extraction of mandibular third molars. MIO measurements are taken using a ruler to measure the distance between the upper and lower central incisors when the participant opens their mouth as wide as possible. Lower values indicate greater trismus.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Friedman JW. The prophylactic extraction of third molars: a public health hazard. Am J Public Health. 2007 Sep;97(9):1554-9. doi: 10.2105/AJPH.2006.100271. Epub 2007 Jul 31. PMID 17666691
- [Background] Meng L, Hua F, Bian Z. Coronavirus Disease 2019 (COVID-19): Emerging and Future Challenges for Dental and Oral Medicine. J Dent Res. 2020 May;99(5):481-487. doi: 10.1177/0022034520914246. Epub 2020 Mar 12. PMID 32162995
- [Background] Long RH, Ward TD, Pruett ME, Coleman JF, Plaisance MC Jr. Modifications of emergency dental clinic protocols to combat COVID-19 transmission. Spec Care Dentist. 2020 May;40(3):219-226. doi: 10.1111/scd.12472. Epub 2020 May 24. PMID 32447777
- [Background] Holland IS, Stassen LF. Bilateral block: is it safe and more efficient during removal of third molars? Br J Oral Maxillofac Surg. 1996 Jun;34(3):243-7. doi: 10.1016/s0266-4356(96)90278-8. PMID 8818259
- [Background] Deepti C, Rehan HS, Mehra P. Changes in quality of life after surgical removal of impacted mandibular third molar teeth. J Maxillofac Oral Surg. 2009 Sep;8(3):257-60. doi: 10.1007/s12663-009-0063-2. Epub 2009 Nov 21. PMID 23139521
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] College C, Feigal R, Wandera A, Strange M. Bilateral versus unilateral mandibular block anesthesia in a pediatric population. Pediatr Dent. 2000 Nov-Dec;22(6):453-7. PMID 11132502
- [Background] Coulthard P, Bailey E, Esposito M, Furness S, Renton TF, Worthington HV. Surgical techniques for the removal of mandibular wisdom teeth. Cochrane Database Syst Rev. 2014 Jul 29;(7):CD004345. doi: 10.1002/14651858.CD004345.pub2. PMID 25069437